CLINICAL TRIAL: NCT02814591
Title: Development of a Novel, Safe Method for the Non-invasive Assessment of Human Bone Quality, In Vivo, Using Spatially Offset Raman Spectroscopy
Brief Title: Development of a Non-invasive Assessment of Human Bone Quality Using Spatially Offset Raman Spectroscopy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: Royal National Orthopaedic Hospital NHS Trust (Other); Science & Technology Facilities Council (Unknown)
Responsible Party: Sponsor
Other Study IDs: 09/0423
Record Dates: First submitted 2016-05-16; First posted 2016-06-28 (Estimated); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Osteoarthritis; Osteoporosis; Osteogenesis Imperfecta; Rickets / Osteomalacia; Bone Infection
MeSH Terms: conditions — Osteoarthritis; Osteoporosis; Osteogenesis Imperfecta; Rickets; Osteomalacia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- Cohort 1: Controls: 40 volunteers free from bone disease. No family histroy of osteogenesis imperfecta (OI). No history of non-accidental fracture. No history of osteoarthritis (OA) or clinical manifestations of disease. No clinical features of OI, OA or osteoporosis (OP). Normal haemoatology and biochemical blood screen. Controls will be gender and age matched (within five years) to the disease cohort patients. Children and adults both required.
  Interventions: Device: spatially offset Raman spectrometer (SORS)
- Cohort 2: Patients with ostegenesis imperfecta (OI).: 40 patients with OI. Patients must have been clinically diagnosed with OI. Participants will be identified form the Royal National Orthopaedic Hospital, Metabolic Unit database. Bone mineral density (BMD) confirmed with DXA.
  Interventions: Device: spatially offset Raman spectrometer (SORS)
- Cohort 3: Patients with osteoarthritis (OA): 40 patients with OA. Patients must have been clinically diagnosed with OA. Participants will be identified from the Royal National Orthopaedic Hospital, Metabolic Unit database.
  Interventions: Device: spatially offset Raman spectrometer (SORS)
- Cohort 4: Patients with osteoporosis (OI): 40 patients with OI receiving treatment with bisphosphonates. Patients must have been clinically diagnosed with OI and bisphosphonates prescribed as a course of treatment. 20 Adults and 20 Children. Where possible participants will be identified from the Royal National Orthopaedic Hospital (RNOH), Metabolic Unit Database; if not from the RNOH then diagnosis will be otherwise confirmed.
  Interventions: Device: spatially offset Raman spectrometer (SORS)
- Cohort 5: Patients with osteoporosis (OP) (2 treatment groups): Patients must have been clinically diagnosed with OP. The first group will have been prescribed with bisphosphonate anti-resorptive treatment; the second with anabolic agents. Where possible participants will be identified from the Royal National Orthopaedic Hospital (RNOH), Metabolic Unit Database; if not from the RNOH then diagnosis will be otherwise confirmed. Bone mineral density (BMD) will be confirmed with DXA. Where possible measurements will be acquired prior to the start of treatment and then up to 4 follow up visits at flexible time points to allow scheduling to coincide with hospital appointments. Minimum time between vistis should be 2 months.
  Interventions: Device: spatially offset Raman spectrometer (SORS)
- Cohort 6: Patients with rickets and osteomalacia: 10-15 participants with rickets and 10-15 participants with osteomalacia. Patients must have been clinically diagnosed with rickets/osteomalacia. Blood tests for 25-hydroxyvitamin D should be less than or equal to 25 nmol/L. Once participants are on treatment further measurements will be made 6 months afterwards. Participants for rickets and osteomalacia groups will be recruited to give a total of 10 complete sets of data per group.
  Interventions: Device: spatially offset Raman spectrometer (SORS)
- Cohort 7: 5 patients with suspected bone infection.: Participants will have been diagnosed at RNOH with a suspected bone infection. Participants will be scanned around the localised area of suspected infection. Participants may have 1 or 2 vists; the latter to take place after all infection has cleared up. This is not subject to a fixed time frame.
  Interventions: Device: spatially offset Raman spectrometer (SORS)

INTERVENTIONS:
Device: spatially offset Raman spectrometer (SORS) — Raman spectra will be collected non-invasively from patients using a lower power 830 nm laser. A probe is brought into gentle contact with the patients skin and measurements taken. The laser power has a pre-defined safe threshold of 30 mW into a 3.5 mm diameter aperture. Built in device safety features prevent this threshold from being exceeded. The probe that comes into patient contact is suitable for disinfecting.

SUMMARY:
In this study spatially offset Raman spectroscopy (SORS), which allows the collection of Raman spectra through turbid media, is being applied to collect Raman spectra of bone. The principal aim to find ways to use Raman spectroscopy to assess bone quality in vivo.

ELIGIBILITY:
INCLUSION CRITERIA

Cohort 1: 40 volunteers, free from bone disease:

* Participants must be free from bone disease and not have a family history of OI;
* Participants to be age and sex matched with OP participants may be recruited among individuals attending the RNOH Metabolic Unit for DXA scanning, who are shown to have normal bone density T score> -2.5;
* No history of non-accidental fracture;
* No history of OA or clinical manifestations of disease;
* No clinical features of OI;
* Controls will be sex and age matched (within five years) to the disease cohort patients.
* Children and adults both required

Cohort 2: 40 patients with OI:

* Patients must have been clinically diagnosed with OI;
* Where possible participants will be identified from the Royal National Orthopaedic Hospital, Metabolic Unit database; if not from RNOH then diagnosis will be otherwise confirmed

Cohort 3: 40 patients with OA:

* Patients must have been clinically diagnosed with OA;
* Participants will be identified from the Royal National Orthopaedic Hospital, Metabolic Unit database; if not from RNOH then diagnosis will be otherwise confirmed

Cohort 4: 40 patients with OI, receiving treatment with bisphosphonates:

* Patients must have been clinically diagnosed with OI and bisphosphonates prescribed as a course of treatment;
* 20 Adults and 20 children
* Where possible participants will be identified from the Royal National Orthopaedic Hospital, Metabolic Unit database; if not from RNOH then diagnosis will be otherwise confirmed
* Where possible measurements will be acquired prior to the start of treatment and then for up to 4 follow up visits at flexible time points to allow scheduling to coincide with hospital appointments. The minimum time between visits should be 2 months.

Cohort 5: 2x 30 patients with OP (two treatment groups):

* Patients must have been clinically diagnosed with OP;
* The first cohort will have been prescribed with bisphosphonate anti-resorptive treatment; the second with anabolic agents. Where treatment has ceased but remains active (long-acting), potential participants may be included at Dr. Keen's discretion.
* Where possible participants will be identified from the Royal National Orthopaedic Hospital, Metabolic Unit database; if not from RNOH then diagnosis will be otherwise confirmed
* BMD confirmed with DXA
* Where possible measurements will be acquired prior to the start of treatment and then up to 4 follow up visits at flexible time points to allow scheduling to coincide with hospital appointments. Minimum time between visits should be 2 months.

Cohort 6: 10-15 participants with rickets, 10-15 participants with osteomalacia

* Patients must have been clinically diagnosed with rickets/osteomalacia;
* Blood tests for 25-hydroxyvitamin D should be ≤25 nmol/L
* Once participants are on treatment a further measurement will be made 6 months afterwards
* Participants for rickets and osteomalacia groups will be recruited to give a total of 10 complete sets of data per group

Cohort 7: 5 participants with a suspected bone infection

* Participants will have been diagnosed at RNOH with a suspected bone infection
* Participants will be scanned around the localised area of suspected infection. Measurements may also be taken away from the infection on the same side and the contralateral anatomical location e.g., if infection is suspected at the right knee then we may also scan further down the right leg and the left leg.
* Participants may have 1 or 2 visits; the latter to take place after all infection has cleared up. This is not subject to a fixed time frame.

EXCLUSION CRITERIA In general smokers will be excluded. Ex-smokers will be included only if they gave up smoking a minimum of 5 years ago.

Cohort 1: 40 volunteers, free from bone disease:

* A participant with a history of bone disease or non-accidental fracture
* Clinical features of bone disease

Cohort 2: 40 patients with OI; Cohort 3: 40 patients with OA; Cohort 6: 20 patients with rickets/osteomalacia • Patients with more than 1 type of bone disease

Cohorts 4, 5 and 6: receiving treatment

• Patients who have been advised to stop treatment. If the treatment is a long-acting one (i.e., will remain effective in the body) then the participant may be included.

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Control patients, patients with osteoarthritis, patients with osteoporosis, patients with osteogenesis imperfecta, patients with rickets or osteomalacia, patients with suspected bone infection.
Sampling Method: Non-Probability Sample
Enrollment: 245 (Estimated)
Dates: Start 2011-10; Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
SORS Raman spectral fingerprint for bone disease types and changes over time | SORS Raman spectral features will be evaluated using a variety of multi-variate analytical tools e.g. BTEM at time zero and a repeat measure within a year.
  Individual patient data will be pre-processed and extracted after patient participation visits. As cohorts are filled multivariate classification models will be built to validate disease discrimination and validation of the SORS technique.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Birch, Professor, Principal Investigator — UCL; Panos Gikas, Consultant Rheumatologist, Principal Investigator — Royal National Orthopaedic Hospital NHS Trust (RNOH)

IPD SHARING:
Plan to Share IPD: Undecided